CLINICAL TRIAL: NCT03648528
Title: Randomized Clinical Trial for The Evaluation of The Effects Of Cholecalciferol Supplementation On The Parathyroid Hormone In Hemodialysis Patients
Brief Title: Cholecalciferol Supplementation Effect on Parathyroid Hormone in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cooperativa Asistencia Sindicato Médico Uruguay (Other)
Responsible Party: Principal Investigator, Laura Sola, Principal Investigator, Cooperativa Asistencia Sindicato Médico Uruguay
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014/004
Record Dates: First submitted 2018-08-10; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Vitamin D Deficiency; Hemodialysis Patient
Keywords: Vitamin D Deficiency; hyperparathyroidism; hemodialysis
MeSH Terms: conditions — Vitamin D Deficiency; Hyperparathyroidism | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Randomized, double blind clinical trial in two arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Bottles filled with cholecalciferol or placebo pills by the drug company (Celsius) and named after randomization by the pharmacist and delivered to the dialysis unit to be administrated by the nurses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cholecaciferol (Experimental): one 5000 IU tablet of 25VD taken during dialysis (3 pills per week) for a period of 12 weeks
  Interventions: Drug: cholecalciferol
- placebo (Placebo Comparator): one tablet of placebo taken during dialysis (3 pills per week) for a period of 12 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cholecalciferol
  Arms: cholecaciferol
Drug: placebo
  Arms: placebo

SUMMARY:
Introduction. Vitamin D regulates mineral metabolism. Its deficiency has been associated with diabetes, cancer and increased mortality. 25OH vitamin D (25VD) is stable and suitable for the evaluation of vitamin D sufficiency.

The aim of the study is to evaluate whether cholecalciferol supplementation for a period of 12 weeks can normalize decreased 25VD levels and reduce increased parathormone (iPTH) in hemodialysis (HD) patients with a vitamin D deficiency. Secondary aims: to evaluate decrease in inflammation, anemia or use of erythropoietin.

Design. Randomized, double blind clinical trial in two arms of HD patients with 25OH Vitamin D deficiency and secondary hyperparathyroidism, for a period of 12 weeks.

Population. Patients over 18 years of age on HD for more than 3 months and levels of 25VD < 30 ng / ml and iPTH >300 ng/ml , who sign a consent form. Randomization will be achieved by using a table of random numbers at the pharmacy, and neither doctors nor patients will know which group they have been assigned to.

Treatment. Supplementation will consist of one 5000 IU cholecalciferol tablet or placebo during dialysis for a period of 12 weeks.

Monthly monitoring will include: haemoglobin (g/dl), Calcium (mg/dl), Phosphorous (mg/dl), PTH (ng/ml), epo dose (IU/kg/week), epo resistance (IU/kg/week/g Hb).

At the beginning and end of the study the following will be measured: alkaline Phosphatase (IU/ml), PCR (mg/L), 25VD (ng/ml), ferritin (ng/ml) and transferrin saturation, quality of life (SF36).

During the study, doses of calcitrol or paricalcitol will not be modified. The study will be discontinued if calcemia ≥ 10.5 mg/dL is detected on two occasions.

Size of sample is estimated at 120 patients for a PTH decrease of 20% in 35% of patients in group treated (assuming 15% follow-up losses). Analysis will be done for Intention to treat for the primary outcome.

Ethical aspects: Authorization has been obtained from the Ethics Committee of the institution as regards Good Clinical Practices, Helsinki Declaration and national regulations. The trial will be registered at the Ministry of Health.

DETAILED DESCRIPTION:
Introduction. Vitamin D regulates mineral metabolism. Its deficiency has been associated with diabetes, cancer and increased mortality. 25OH vitamin D (25VD) is stable and suitable for the evaluation of vitamin D sufficiency.

The aim of the study is to evaluate whether cholecalciferol supplementation for a period of 12 weeks can normalize decreased levels of 25VD and reduce increased parathormone (iPTH) in hemodialysis (HD) patients with a vitamin D deficiency. Secondary aims: to evaluate decrease in inflammation, anemia or use of erythropoietin (epo).

Design. Randomized, double blind clinical trial in two arms of HD patients with 25VD deficiency and secondary hyperparathyroidism, one arm to be treated with cholecalciferol supplementation and the other with a placebo, for a period of 12 weeks.

Population. Patients over 18 years of age on HD for more than 3 months and levels of 25VD < 30 ng / ml and iPTH >300 ng/ml , who sign a consent form. Once their consent has been obtained, iPTH and 25VD levels will be measured. Randomization will be achieved by using a table of random numbers at the pharmacy, and neither doctors nor patients will know which group they have been assigned to.

Treatment. Supplementation will consist of three 5000 IU cholecalciferol tablets or placebo postdialysis per week during dialysis for a period of 12 weeks.

Monthly monitoring will include: haemoglobin (g/dl), Calcium (mg/dl), Phosphorous (mg/dl), iPTH (ng/ml), epo dose (IU/kg/week), epo resistance (IU/kg/week/g Hb).

At the beginning and end of the study the following will be measured: alkaline Phosphatase (IU/ml), C reactive protein (mg/L), 25VD (ng/ml), ferritin (ng/ml) and transferrin saturation, quality of life (SF36).

During the study, doses of calcitrol or paricalcitol will not be modified. The study will be discontinued if calcemia ≥ 10.5 mg/dL is detected on two occasions.

Size of sample is estimated at 120 patients for a iPTH decrease of 20% in 35% of patients in group treated (assuming 15% follow-up losses). Analysis will be done for Intention to treat for the primary outcome.

Ethical aspects: Authorization has been obtained from the Ethics Committee of the institution as regards Good Clinical Practices, Helsinki Declaration and national regulations. The trial was registered at the Ministry of Health.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* signed informed consent form
* ESRD with regular dialysis treatment for at least 3 months
* levels of 25VD < 30 ng / ml
* levels of iPTH >300 ng/ml,
* stable doses of calcitrol or paricalcitol over the last 30 days.

Exclusion Criteria:

* Congestive heart failure class III or IV
* unstable angina or myocardial infarction or stroke during the previous 3 months
* active malignant neoplasm
* use of any trial medication
* life expectancy lower than 6 months
* corrected calcemia ≥ 10.5 in the 2 months prior to recruitment
* intake of cholecalciferol or ergocalciferol in the 2 months prior to recruitment
* prospective move to another city or transfer to PD in the following 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
20 % Change in iPTH levels | 12 weeks
  20% change on final iPTH level
normalization of 25VD levels | 12 weeks
  % of patients achieving normal 25VD levels

SECONDARY OUTCOMES:
change of 0.5 g/dL on Hb level or 10% change in erythropoietin dose | 12 weeks
  change of 0.5 g/dL on Hb level or 10% change in erythropoietin dose

DOCUMENTS (2):
  • Study Protocol (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT03648528/Prot_000.pdf
  • Informed Consent Form (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT03648528/ICF_001.pdf